CLINICAL TRIAL: NCT01492088
Title: A Phase 1/2 Study of Brentuximab Vedotin (SGN-35) in Pediatric Patients With Relapsed or Refractory Systemic Anaplastic Large-Cell Lymphoma or Hodgkin Lymphoma
Brief Title: Study of Brentuximab Vedotin (SGN-35) in Pediatric Participants With Relapsed or Refractory (r/r) Systemic Anaplastic Large-Cell Lymphoma or Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C25002; 2011-001240-29 (EudraCT Number); U1111-1158-2613 (Registry Identifier: WHO); 133300410A0384 (Registry Identifier: RNEC); NL38209.078.11 (Registry Identifier: CCMO)
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Relapsed or Refractory Hodgkin Lymphoma; Relapsed or Refractory Anaplastic Large-cell Lymphoma
Keywords: Pediatric; Lymphoma; Hodgkin; Anaplastic Large-cell; Relapsed; Refractory; Drug therapy
MeSH Terms: conditions — Recurrence; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Lymphoma | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brentuximab vedotin: Phase 1 (Experimental): Brentuximab vedotin 1.4 mg/kg, 30-minute IV infusion, Day 1 of every 21-day cycle, until there was evidence of disease progression or unacceptable toxicity. Dose was escalated up to 1.8 mg/kg using a 3 + 3 dose escalation design to determine a maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) depending upon the dose limiting toxicity (DLT).
  Interventions: Drug: Brentuximab vedotin
- Brentuximab vedotin: Phase 2 (Experimental): Brentuximab vedotin 1.8 mg/kg, 30-minute IV infusion, Day 1 of every 21-day cycle, until there is evidence of disease progression or unacceptable toxicity (Up to 16 cycles). Treatment with brentuximab vedotin beyond 16 cycles was permitted at the joint discretion of the sponsor and the investigator for those participants experiencing continued clinical benefit.
  Interventions: Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Brentuximab vedotin — Brentuximab vedotin IV infusion
  Other Names: SGN-35; ADCETRIS

SUMMARY:
The purpose of this study is to assess the safety and pharmacokinetics, and determine the pediatric maximum tolerated dose and/or or recommended phase 2 dose of brentuximab vedotin.

DETAILED DESCRIPTION:
The drug being tested in this study is called brentuximab vedotin. Brentuximab vedotin is being tested to treat children who have relapsed or refractory (r/r) anaplastic large-cell lymphoma (sALCL) or Hodgkin lymphoma (HL). This study will look at the maximum tolerated dose and/or recommended phase 2 dose, safety and pharmacokinetics of brentuximab vedotin along with overall response of people who took brentuximab vedotin.

The study enrolled 36 patients. In the phase 1 portion of the study, 12 participants were enrolled to receive brentuximab vedotin 1.4-1.8 mg/kg, 30-minute IV infusion, Day 1 of every 21-day cycle, until there was evidence of disease progression or unacceptable toxicity.

Once the maximum tolerated dose and/or recommended phase 2 dose and pharmacokinetics of brentuximab vedotin was reached, participants were enrolled by diagnosis into two phase 2 study arms: relapsed or refractory sALCL or relapsed or refractory HL and received brentuximab vedotin 1.8 mg/kg as 30-minute IV on Day 1 of every 21-day cycle for up to 16 cycles. One participant received a maximum of 20 cycles at the joint discretion of the sponsor and the investigator for continued clinical benefit.

This multicenter trial is being conducted worldwide. The overall time to participate in this study is approximately 5 years. Participants made multiple visits to the clinic, and were contacted by telephone every 12 weeks for 12 months after the end of treatment (EOT) for progression free survival and then every 6 months until death, study closure, or 2 years after enrollment of the last participant for overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 2 to <18 years (5 to <18 years for Hodgkin lymphoma [HL])
* Diagnosis of systemic anaplastic large-cell lymphoma (sALCL), or HL for which standard, curative, life-prolonging, or palliative treatment does not exist or is no longer effective
* Participants with sALCL must have documented anaplastic lymphoma kinase (ALK) status and must be beyond first remission or refractory to front-line chemotherapy
* Participants diagnosed with any relapsed or refractory CD30+ hematologic malignancy (e.g., primary mediastinal B-cell lymphoma) may be included in phase 1 of the study
* Participants with HL must be in their second of later relapse, have failed systemic chemotherapy either as induction therapy for advanced stage disease or salvage therapy, and were ineligible for, refused, or previously received a stem cell transplant
* Performance score ≥ 60 from Lansky Play Performance Scale if ≤16 years
* Negative pregnancy test
* Fertile Participants must use 2 effective methods of contraception prior to and through 6 months after the last dose of the study drug

Exclusion Criteria:

* Current diagnosis of primary cutaneous ALCL (those with systemic ALCL are eligible)
* Received an allogeneic stem cell transplant <3 months prior to the first dose of study medication, or presence of polymerase chain reaction (PCR)-detectable cytomegalovirus (CMV) in any post-allogeneic transplant participant
* Receiving immunosuppressive therapy
* Receiving systemic therapy for chronic graft-versus-host disease (topical therapy is allowed)
* Previous treatment with any anti-CD30 antibody
* Therapeutic monoclonal antibody use within the longer of 6 weeks or 5 plasma half-lives
* Systemic cardiac disease that would, in the opinion of the investigator or medical monitor, interfere with assessment of efficacy or safety of the drug
* History of another primary malignancy not in remission for at least 3 years (the following are exempt from the 3-year limit: nonmelanoma skin cancer and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Pap smear)
* Known active cerebral/meningeal disease, including signs or symptoms of progressive multifocal leukoencephalopathy (PML) or any history of PML
* History of cirrhosis
* Active systemic viral, bacterial, or fungal infection requiring antimicrobial, antiviral therapy or antifungal therapy within 2 weeks prior to the first dose of study drug (routine antimicrobial prophylaxis is acceptable)
* Concurrent therapy with other anti-neoplastic or experimental agents
* Systemic corticosteroid therapy <7 days prior to first dose of the study medication
* Any serious underlying medical condition that, in the opinion of the investigator or medical monitor, would impair their ability to receive or tolerate the planned treatment
* Known hypersensitivity to recombinant proteins, murine proteins, or any excipient contained in the drug formulation
* Received nitrogen mustard agents, melphalan, or BCNU therapy within 6 weeks prior to the first study dose
* Prior autologous hematopoietic stem cell infusion <4 weeks prior to first study dose
* Grade 2 or greater unresolved toxicity from prior antineoplastic therapy
* Grade 2 or greater peripheral neuropathy
* Female participants who are both lactating and breastfeeding, or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before the first dose of study drug
* Received local palliative radiation therapy <14 days prior to the first dose of study medication
* Received radiation therapy to more than 25% of the bone marrow-containing spaces < 84 days prior to first dose of study medication
* Received a strong or listed moderate inhibitor of CYP3A4 <2 weeks prior to first study dose
* Participants must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2012-04-16 (Actual); Primary Completion 2016-10-12 (Actual); Study Completion 2018-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (18):
- United States (4):
  - Aurora, Colorado
  - Kansas City, Missouri
  - New York, New York
  - Houston, Texas
- France (3):
  - Bordeaux
  - Lyon
  - Paris
- Germany (5):
  - Berlin
  - Frankfurt
  - Giessen
  - Halle
  - Münster
- Italy (2):
  - Padua
  - Roma
- Mexico City, Mexico
- Rotterdam, Netherlands
- Barcelona, Spain
- London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Result] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Derived] Suri A, Mould DR, Song G, Kinley J, Venkatakrishnan K. Population Pharmacokinetics of Brentuximab Vedotin in Adult and Pediatric Patients With Relapsed/Refractory Hematologic Malignancies: Model-Informed Hypothesis Generation for Pediatric Dosing Regimens. J Clin Pharmacol. 2020 Dec;60(12):1585-1597. doi: 10.1002/jcph.1682. Epub 2020 Jun 28. PMID 32596842
- [Derived] Locatelli F, Mauz-Koerholz C, Neville K, Llort A, Beishuizen A, Daw S, Pillon M, Aladjidi N, Klingebiel T, Landman-Parker J, Medina-Sanson A, August K, Sachs J, Hoffman K, Kinley J, Song S, Song G, Zhang S, Suri A, Gore L. Brentuximab vedotin for paediatric relapsed or refractory Hodgkin's lymphoma and anaplastic large-cell lymphoma: a multicentre, open-label, phase 1/2 study. Lancet Haematol. 2018 Oct;5(10):e450-e461. doi: 10.1016/S2352-3026(18)30153-4. PMID 30290902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 investigative sites in United States, France, Germany, Netherlands, United Kingdom, Italy, Spain and Mexico from 16-April-2012 to 12-April-2018.
Pre-assignment Details: Participants with diagnosis of relapsed or refractory (r/r) sALCL/HL were enrolled to receive brentuximab vedotin 1.4-1.8 mg/kg, intravenous infusion on Day 1 of every 21-day cycle for up to 16 cycles. Treatment beyond 16 cycles was permitted at joint discretion of sponsor and investigator for participants experiencing continued clinical benefit.
Groups:
- Brentuximab Vedotin 1.4 mg/kg: Phase 1: Brentuximab vedotin 1.4 mg/kg, 30-minute IV infusion, Day 1 of every 21-day cycle, until there was evidence of disease progression or unacceptable toxicity.
- Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only: Participants with r/r HL received brentuximab vedotin 1.8 mg/kg, 30-minute IV infusion, Day 1 of every 21-day cycle until there was evidence of disease progression or unacceptable toxicity (Up to 16 cycles). Treatment with brentuximab vedotin beyond 16 cycles was permitted at the joint discretion of the sponsor and the investigator for those participants experiencing continued clinical benefit.
- Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only: Participants with r/r systemic anaplastic large-cell lymphoma (sALCL) received brentuximab vedotin 1.8 mg/kg, 30-minute IV infusion, Day 1 of every 21-day cycle until there was evidence of disease progression or unacceptable toxicity (Up to 16 cycles). Treatment with brentuximab vedotin beyond 16 cycles was permitted at the joint discretion of the sponsor and the investigator for those participants experiencing continued clinical benefit.
Period: Overall Study
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only
Started | 3 | 16 | 17
Completed | 0 | 2 | 3
Not Completed | 3 | 14 | 14
Not completed — Withdrawal by Patient | 0 | 2 | 0
Not completed — Death | 1 | 6 | 2
Not completed — Completed Post Treatment Followup (PTFU) | 2 | 0 | 1
Not completed — Alive at Last Follow-up | 0 | 6 | 11

BASELINE CHARACTERISTICS:
Population: Safety population is defined as participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only | Total
Number analyzed (Participants) | 3 | 16 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.15) | 14.5 (2.68) | 11.5 (3.18) | 13.1 (3.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 3 | 11
  Male | 2 | 9 | 14 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 4 | 4
  Not Hispanic or Latino | 3 | 14 | 12 | 29
  Unknown or Not Reported | 0 | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 13 | 16 | 31
  Asian | 1 | 0 | 1 | 2
  Other | 0 | 2 | 0 | 2
  Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 1 | 4
  France | 0 | 2 | 0 | 2
  Germany | 0 | 4 | 1 | 5
  Netherlands | 0 | 1 | 2 | 3
  United Kingdom | 0 | 1 | 2 | 3
  Italy | 1 | 7 | 6 | 14
  Spain | 0 | 0 | 4 | 4
  Mexico | 0 | 0 | 1 | 1
Height [Mean (Standard Deviation); unit: cm] | 167.17 (10.865) | 165.31 (14.350) | 149.54 (17.783) | 158.02 (17.493)
Weight [Mean (Standard Deviation); unit: kg] | 53.10 (9.924) | 57.85 (17.539) | 42.16 (15.162) | 50.04 (17.361)
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.562 (0.0967) | 1.617 (0.2938) | 1.313 (0.3103) | 1.469 (0.3228)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) (Phase 1)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A Serious Adverse Event (SAE) is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. AE severity was graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.
Time Frame: From the first dose through 30 days after the last dose of study medication (Up to 15 months)
Population: Safety population is defined as all participants who received at least 1 dose of study drug. Participants enrolled in Phase 1 of study were evaluated for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Brentuximab Vedotin 1.8 mg/kg: Phase 1: Brentuximab vedotin 1.8 mg/kg, 30-minute IV infusion, Day 1 of every 21-day cycle until there was evidence of disease progression or unacceptable toxicity (Up to 16 cycles). Treatment with brentuximab vedotin beyond 16 cycles was permitted at the joint discretion of the sponsor and the investigator for those participants experiencing continued clinical benefit.
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1
Number analyzed (Participants) | 3 | 9
Participants
  TEAE | 3 | 9
  SAE | 0 | 4

2. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Values Reported as AEs (Phase 1)
Description: Abnormal clinical laboratory values (serum chemistry and hematology) were reported as AEs if they were considered by the investigator to be a clinically significant change from Baseline or led to premature discontinuation of study treatment, dose modification, or other therapeutic intervention.
Time Frame: From the first dose through 30 days after the last dose of study medication (Up to 15 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1
Number analyzed (Participants) | 3 | 9
Participants
  Gamma-glutamyltransferase increased | 0 | 1
  Transaminases increased | 0 | 1
  Lymphocyte count decreased | 1 | 1
  Neutrophil count decreased | 0 | 1
  Blood bicarbonate decreased | 0 | 1
  Weight decreased | 0 | 1
  Hypocalaemia | 0 | 2
  Hyperuricaemia | 0 | 1

3. Primary Outcome: Number of Participants With Clinically Significant Vital Signs Values Reported as AEs (Phase 1)
Description: Vital signs measurements included supine (after 3-5 minutes in this position) and standing (after 3-5 minutes in this position) measurements of diastolic and systolic blood pressure, heart rate, and oral temperature.
Time Frame: From the first dose through 30 days after the last dose of study medication (Up to 15 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Brentuximab Vedotin 1.8 mg/kg: Phase 1: Brentuximab vedotin 1.8 mg/kg, 30-minute IV infusion, Day 1 of every 21-day cycle starting from Cycle 2 until there was evidence of disease progression or unacceptable toxicity (Up to 16 cycles). Treatment with brentuximab vedotin beyond 16 cycles was permitted at the joint discretion of the sponsor and the investigator for those participants experiencing continued clinical benefit.
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1
Number analyzed (Participants) | 3 | 9
Participants | 0 | 0

4. Primary Outcome: Antibody-drug Conjugate (ADC) Serum Concentrations (Phase 1)
Description: Blood samples were collected and tested for serum concentrations of brentuximab vedotin antibody-drug conjugate.
Time Frame: Cycle 1 and 8 pre-dose and 5 minutes, 24, 48, 96 and 312 hours post-dose; Cycle 2 pre-dose, 5 minutes and 24, 48 and 96 hours post-dose; Cycle 3 to 16 pre-dose and 5 minutes post-dose
Population: Data for this outcome measure was not summarized for Phase 1 participants only, data was summarized together for Phase 1 and 2 participants in brentuximab 1.4 mg/kg and 1.8 mg/kg arms groups. Data has been presented in OM 19.
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Serum Concentration of Total Antibodies (Conjugated and Unconjugated) (Phase 1)
Description: Blood samples were collected and tested for conjugated and unconjugated antibodies.
Time Frame: as for outcome 4
Population: Data for this outcome measure was not summarized for Phase 1 participants only, data was summarized together for Phase 1 and 2 participants in brentuximab 1.4 mg/kg and 1.8 mg/kg arms groups. Data has been presented in OM 20.
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Monomethyl Auristatin E (MMAE) Plasma Concentrations (Phase 1)
Description: Blood samples were collected and tested for MMAE plasma concentrations.
Time Frame: as for outcome 4
Population: Data for this outcome measure was not summarized for Phase 1 participants only, data was summarized together for Phase 1 and 2 participants in brentuximab 1.4 mg/kg and 1.8 mg/kg arms groups. Data has been presented in OM 21.
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Overall Response Rate (ORR) (Phase 1 and 2)
Description: Overall response rate is defined as the percentage of participants with complete remission (CR) or partial remission (PR) as assessed by an independent review facility (IRF) using International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma. CR is defined as the disappearance of all evidence of disease and PR is defined as regression of measurable disease and no new sites.
Time Frame: Cycles 2, 4, 7, 10, 13 and 16 (21-day cycles) until disease progression, death or end of treatment (EOT) (Up to 15 months)
Population: Response-evaluable population included participants who received at least 1 dose of study drug, have measurable disease at baseline, and 1 postbaseline disease assessment. Data was summarized together for Phase 1 and 2 participants in brentuximab 1.8 mg/kg arm group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only: Participants with r/r Hodgkin Lymphoma (HL) received brentuximab vedotin 1.8 mg/kg, 30-minute IV infusion, Day 1 of every 21-day cycle until there was evidence of disease progression or unacceptable toxicity (Up to 16 cycles). Treatment with brentuximab vedotin beyond 16 cycles was permitted at the joint discretion of the sponsor and the investigator for those participants experiencing continued clinical benefit.
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only
Number analyzed (Participants) | 3 | 15 | 17
percentage of participants | 0 [0 to 71] | 47 [21 to 73] | 53 [28 to 77]

8. Secondary Outcome: Number of Participants With Antitherapeutic Antibodies (ATA) and Neutralizing ATA (nATA) (Phase 1 and 2)
Description: Blood samples were collected to assess the immunogenicity of brentuximab vedotin (ATA and nATA development) using a laboratory test. ATA-positive samples were further characterized as transiently ATA positive (defined as 1 or 2 post-Baseline ATA-positive responses), persistently ATA positive (defined as more than 2 post-Baseline ATA positive responses), and nATA positive or negative.
Time Frame: Baseline up to EOT (Up to 15 months)
Population: Participants from the Safety Population, all enrolled participants who received at least one dose of brentuximab vedotin, with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only
Number analyzed (Participants) | 3 | 16 | 17
Participants
  ATA status: Transiently positive | 1 | 4 | 7
  ATA status: Persistently positive | 0 | 2 | 0
  nATA status: Positive | 0 | 5 | 4

9. Secondary Outcome: Overall Response Rate (ORR) (Phase 1)
Description: Overall response rate is defined as the percentage of participants with CR or PR as assessed by an IRF using IWG Revised Response Criteria for Malignant Lymphoma. CR is defined as the disappearance of all evidence of disease and PR is defined as regression of measurable disease and no new sites.
Time Frame: Cycles 2, 4, 7, 10, 13 and 16 (21-day cycles) until disease progression, death or EOT (Up to 15 months)
Population: Response-evaluable population included participants who received at least 1 dose of study drug, have measurable disease at baseline, and 1 postbaseline disease assessment. Participants enrolled in Phase 1 of the study were evaluated for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1
Number analyzed (Participants) | 3 | 8
percentage of participants | 0 [0 to 71] | 63 [24 to 91]

10. Secondary Outcome: Time to Progression (TTP) (Phase 1 and 2)
Description: TTP is defined as the time in months from first dose until the first subsequent documentation of objective tumor progression. Progressive disease (PD) is defined as any new lesion or increase by ≥50% of previously involved sites from nadir.
Time Frame: Cycles 2, 4, 7, 10, 13 and 16 (21-day cycles) until disease progression, death or EOT and then every 12 weeks for 12 months after EOT, until disease progression, or death (Up to 27 months)
Population: Safety population is defined as all participants who received at least 1 dose of study drug. TTP was censored on last radiological assessment of measured lesions documenting absence of PD for participants who did not have tumor progression.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only
Number analyzed (Participants) | 3 | 16 | 17
months | 2.7 [1.4 to 2.8] | 4.8 [1.2 to NA] — Upper limit of CI was not reached due to low number of participants with events. | 6.2 [2.8 to NA] — Upper limit of CI was not reached due to low number of participants with events.

11. Secondary Outcome: Time to Response (Phase 1 and 2)
Description: Time to response is defined as the time in months from the first dose of study treatment until the date of the first assessment of confirmed CR or PR. as assessed by an IRF using IWG revised response criteria for malignant lymphoma. CR is defined as the disappearance of all evidence of disease and PR is defined as regression of measurable disease and no new sites.
Time Frame: Cycles 2, 4, 7, 10, 13 and 16 (21-day cycles) until disease progression, death or EOT (Up to 15 months)
Population: Response-evaluable population included participants who received at least 1 dose of study drug, have measurable disease at baseline, and 1 postbaseline disease assessment. Time to response was censored on the last radiological assessment of measured lesions documenting absence of CR or PR for participants who did not have CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only
Number analyzed (Participants) | 3 | 15 | 17
months | NA [NA to NA] — Median was not reached as no participant had response. | 2.7 [1.3 to NA] — Upper limit of CI was not reached due to low number of participants with events. | 1.5 [1.2 to NA] — Upper limit of CI was not reached due to low number of participants with events.

12. Secondary Outcome: Duration of Response (DOR) (Phase 1 and 2)
Description: DOR is defined as the time in months from the date of first documentation of a CR or PR to the date of first documentation of tumor progression or PD per IRF assessment according to IWG criteria or to death due to any cause, whichever comes first. CR is defined as the disappearance of all evidence of disease and PD is defined as any new lesion or increase by >50% of previously involved sites from nadir.
Time Frame: Cycles 2, 4, 7, 10, 13 and 16 (21-day cycles) until disease progression, death or EOT and then every 12 weeks for 12 months after EOT, until disease progression, or death or end of study (Up to 72 months)
Population: Participants with response from the Safety Population, all enrolled participants who received at least one dose of brentuximab vedotin, with data available for analysis. Duration of response was censored at last observation documenting absence of PD for participants who did not have tumor progression.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only
Number analyzed (Participants) | 0 | 7 | 9
months |  | NA [2.2 to NA] — Median and upper limit of CI was not reached due to low number of participants with events. | 30.3 [3.4 to 30.3]

13. Secondary Outcome: Event Free Survival (EFS) (Phase 1 and 2)
Description: EFS is defined as the time in months from first dose until any cause of treatment failure: disease progression, premature discontinuation of treatment for any reason, or death due to any cause, whichever occurs first. PD is defined as any new lesion or increase by >50% of previously involved sites from nadir.
Time Frame: as for outcome 10
Population: Safety population is defined as all participants who received at least 1 dose of study drug. EFS was censored on the last follow-up date if none of the above events occur during the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only
Number analyzed (Participants) | 3 | 16 | 17
months | 2.7 [1.4 to 2.8] | 2.1 [1.2 to 4.8] | 4.8 [2.8 to 7.4]

14. Secondary Outcome: Progression Free Survival (PFS) (Phase 1 and 2)
Description: PFS is defined as time in months from start of study treatment to first documentation of objective tumor progression per IRF assessment or up to death due to any cause, whichever occurs first. PD is defined as any new lesion or increase by >50% of previously involved sites from nadir.
Time Frame: as for outcome 12
Population: Safety population is defined as all participants who received at least 1 dose of study drug. PFS was censored on the day following the date of last radiological assessment of measured lesions documenting absence of PD for participants who did not have tumor progression.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only
Number analyzed (Participants) | 3 | 16 | 17
months | 2.7 [1.4 to 2.8] | 3.8 [1.2 to NA] — Upper limit of CI was not reached due to low number of participants with events. | 6.2 [2.8 to 31.5]

15. Secondary Outcome: Overall Survival (OS) (Phase 1 and 2)
Description: OS is the time in months from start of study treatment to date of death due to any cause.
Time Frame: Every 6 months after EOT, until the sooner of death, study closure, or 2 years after enrolment of the last participant (Up to 72 months)
Population: Safety population is defined as all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only
Number analyzed (Participants) | 3 | 16 | 17
months | NA [NA to NA] — Median was not reached due to low number of participants with events. | NA [NA to NA] — Median was not reached due to low number of participants with events. | NA [NA to NA] — Median was not reached due to low number of participants with events.

16. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) (Phase 1 and 2)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A SAE is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. AE severity was graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.
Time Frame: From the first dose through 30 days after the last dose of study medication (up to 15 months)
Population: Safety population is defined as all participants who received at least 1 dose of study drug. Data was summarized together for Phase 1 and 2 participants in brentuximab 1.8 mg/kg arm group.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only
Number analyzed (Participants) | 3 | 16 | 17
Participants
  TEAEs | 3 | 16 | 17
  SAEs | 0 | 7 | 1

17. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Values Reported as AEs (Phase 1 and 2)
Description: as for outcome 2
Time Frame: From the first dose through 30 days after the last dose of study medication (Up to 15 months)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only
Number analyzed (Participants) | 3 | 16 | 17
Participants
  Gamma-glutamyltransferase increased | 0 | 2 | 0
  Alanine aminotransferase increased | 0 | 1 | 0
  Aspartate aminotransferase increased | 0 | 1 | 0
  Transaminases increased | 0 | 1 | 0
  Lymphocyte count decreased | 1 | 0 | 2
  Neutrophil count decreased | 0 | 0 | 2
  White blood cell count decreased | 0 | 0 | 1
  Blood bicarbonate decreased | 0 | 1 | 0
  Weight decreased | 0 | 0 | 1
  C-reactive protein increased | 0 | 1 | 0
  Blood alkaline phosphatase increased | 0 | 1 | 0

18. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Reported as AEs (Phase 1 and 2)
Description: as for outcome 3
Time Frame: From the first dose through 30 days after the last dose of study medication (Up to 15 months)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only
Number analyzed (Participants) | 3 | 16 | 17
Participants | 0 | 0 | 0

19. Secondary Outcome: Antibody-drug Conjugate (ADC) Serum Concentrations (Phase 1 and 2)
Description: Blood samples were collected and tested for serum concentrations of brentuximab vedotin antibody-drug conjugate.
Time Frame: as for outcome 4
Population: PK-evaluable population was defined as participants with sufficient dosing and PK data to reliably estimate PK parameters. Cycle 2 Day 2 values are collected in phase 1 participants only. Here, number analyzed is number of participants assessed at given time-point. Data summarized together for all participants in brentuximab vedotin 1.8 mg/kg arm.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1
Number analyzed (Participants) | 3 | 33
ug/mL
  Cycle 1 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 33
  Cycle 1 Day 1, Pre-Dose |  | NA (NA) — Data was below the limit of quantification.
  Cycle 1 Day 1, 5 Minutes Post-Dose | 23.1 (3.46) | 31.8 (12.4)
  Cycle 1 Day 2, 24 Hours Post-Dose: number analyzed (Participants) | 3 | 32
  Cycle 1 Day 2, 24 Hours Post-Dose | 9.50 (1.73) | 13.0 (5.34)
  Cycle 1 Day 3, 48 Hours Post-Dose: number analyzed (Participants) | 3 | 31
  Cycle 1 Day 3, 48 Hours Post-Dose | 5.67 (0.924) | 12.0 (16.3)
  Cycle 1 Day 5, 96 Hours Post-Dose: number analyzed (Participants) | 3 | 31
  Cycle 1 Day 5, 96 Hours Post-Dose | 3.50 (1.41) | 8.68 (13.4)
  Cycle 1 Day 14, 312 Hours Post-Dose: number analyzed (Participants) | 3 | 31
  Cycle 1 Day 14, 312 Hours Post-Dose | 0.844 (0.309) | 2.19 (3.44)
  Cycle 2 Day 1, Pre-Dose: number analyzed (Participants) | 3 | 32
  Cycle 2 Day 1, Pre-Dose | 0.149 (0.128) | 0.395 (0.322)
  Cycle 2 Day 1, 5-minutes Post-Dose: number analyzed (Participants) | 3 | 30
  Cycle 2 Day 1, 5-minutes Post-Dose | 25.3 (7.56) | 32.9 (9.80)
  Cycle 2 Day 2, 24 Hours Post-Dose: number analyzed (Participants) | 3 | 10
  Cycle 2 Day 2, 24 Hours Post-Dose | 8.80 (6.19) | 10.4 (8.05)
  Cycle 2 Day 3, 48 Hours Post-Dose: number analyzed (Participants) | 3 | 29
  Cycle 2 Day 3, 48 Hours Post-Dose | 3.70 (1.95) | 11.4 (16.8)
  Cycle 2 Day 5, 96 Hours Post-Dose: number analyzed (Participants) | 3 | 27
  Cycle 2 Day 5, 96 Hours Post-Dose | 2.04 (1.26) | 9.61 (17.9)
  Cycle 3 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 26
  Cycle 3 Day 1, Pre-Dose | 0.116 (0.163) | 0.491 (0.387)
  Cycle 3 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 26
  Cycle 3 Day 1, 5 minutes Post-Dose | 23.9 (2.83) | 31.3 (9.79)
  Cycle 4 Day 1, Pre-dose: number analyzed (Participants) | 2 | 21
  Cycle 4 Day 1, Pre-dose | 0.218 (0.271) | 0.691 (0.492)
  Cycle 4 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 21
  Cycle 4 Day 1, 5 minutes Post-Dose | 22.9 (4.60) | 30.0 (12.2)
  Cycle 5 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 21
  Cycle 5 Day 1, Pre-Dose | 0.264 (0.321) | 0.845 (0.564)
  Cycle 5 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 21
  Cycle 5 Day 1, 5 minutes Post-Dose | 22.5 (3.32) | 30.6 (15.1)
  Cycle 6 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 17
  Cycle 6 Day 1, Pre-Dose | 0.312 (0.351) | 1.06 (0.699)
  Cycle 6 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 17
  Cycle 6 Day 1, 5 minutes Post-Dose | 20.3 (4.38) | 33.2 (16.1)
  Cycle 7 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 17
  Cycle 7 Day 1, Pre-Dose | 0.327 (0.337) | 1.04 (0.618)
  Cycle 7 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 17
  Cycle 7 Day 1, 5 minutes Post-Dose | 17.9 (2.40) | 32.3 (15.4)
  Cycle 8 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 14
  Cycle 8 Day 1, Pre-Dose |  | 1.25 (0.565)
  Cycle 8 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 14
  Cycle 8 Day 1, 5 minutes Post-Dose |  | 35.2 (10.5)
  Cycle 8 Day 2, 24 Hours Post-Dose: number analyzed (Participants) | 0 | 13
  Cycle 8 Day 2, 24 Hours Post-Dose |  | 14.0 (4.55)
  Cycle 8 Day 3, 48 Hours Post-Dose: number analyzed (Participants) | 0 | 13
  Cycle 8 Day 3, 48 Hours Post-Dose |  | 9.53 (2.96)
  Cycle 8 Day 5, 96 Hours Post-Dose: number analyzed (Participants) | 0 | 12
  Cycle 8 Day 5, 96 Hours Post-Dose |  | 6.44 (2.35)
  Cycle 8 Day 14, 312 Hours Post-Dose: number analyzed (Participants) | 0 | 13
  Cycle 8 Day 14, 312 Hours Post-Dose |  | 3.30 (4.63)
  Cycle 9 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 14
  Cycle 9 Day 1, Pre-Dose |  | 4.37 (11.7)
  Cycle 9 Day 1, 5 Minutes Post-Dose: number analyzed (Participants) | 0 | 13
  Cycle 9 Day 1, 5 Minutes Post-Dose |  | 29.6 (11.3)
  Cycle 10 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 11
  Cycle 10 Day 1, Pre-Dose |  | 1.20 (0.455)
  Cycle 10 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 12
  Cycle 10 Day 1, 5 minutes Post-Dose |  | 35.7 (9.50)
  Cycle 11 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 8
  Cycle 11 Day 1, Pre-Dose |  | 1.84 (1.57)
  Cycle 11 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 8
  Cycle 11 Day 1, 5 minutes Post-Dose |  | 35.7 (10.8)
  Cycle 12 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 12 Day 1, Pre-Dose |  | 1.47 (0.665)
  Cycle 12 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 6
  Cycle 12 Day 1, 5 minutes Post-Dose |  | 40.0 (10.4)
  Cycle 13 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 13 Day 1, Pre-Dose |  | 6.28 (11.5)
  Cycle 13 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 6
  Cycle 13 Day 1, 5 minutes Post-Dose |  | 33.3 (16.1)
  Cycle 14 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 14 Day 1, Pre-Dose |  | 1.60 (0.600)
  Cycle 14 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 6
  Cycle 14 Day 1, 5 minutes Post-Dose |  | 37.0 (7.92)
  Cycle 15 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 15 Day 1, Pre-Dose |  | 1.48 (0.542)
  Cycle 15 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 6
  Cycle 15 Day 1, 5 minutes Post-Dose |  | 40.3 (10.6)
  Cycle 16 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 16 Day 1, Pre-Dose |  | 1.52 (0.361)
  Cycle 16 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 6
  Cycle 16 Day 1, 5 minutes Post-Dose |  | 41.5 (4.70)

20. Secondary Outcome: Serum Concentration of Total Antibodies (Conjugated and Unconjugated)
Description: Blood samples were collected and tested for conjugated and unconjugated antibodies.
Time Frame: as for outcome 4
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1
Number analyzed (Participants) | 3 | 33
ug/mL
  Cycle 1 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 32
  Cycle 1 Day 1, Pre-Dose | NA (NA) — Data was below the limit of quantification. | NA (NA) — Data was below the limit of quantification.
  Cycle 1 Day 1, 5 Minutes Post-Dose | 26.3 (2.29) | 34.7 (13.4)
  Cycle 1 Day 2, 24 Hours Post-Dose | 16.7 (1.50) | 25.0 (9.59)
  Cycle 1 Day 3, 48 Hours Post-Dose | 12.7 (3.13) | 18.5 (7.57)
  Cycle 1 Day 5, 96 Hours Post-Dose | 8.63 (5.11) | 11.8 (5.02)
  Cycle 1 Day 14, 312 Hours Post-Dose: number analyzed (Participants) | 3 | 32
  Cycle 1 Day 14, 312 Hours Post-Dose | 2.23 (0.833) | 3.50 (1.70)
  Cycle 2 Day 1, Pre-Dose: number analyzed (Participants) | 3 | 32
  Cycle 2 Day 1, Pre-Dose | 0.470 (0.459) | 1.16 (0.825)
  Cycle 2 Day 1, 5-minutes Post-Dose: number analyzed (Participants) | 3 | 31
  Cycle 2 Day 1, 5-minutes Post-Dose | 26.9 (7.98) | 35.6 (12.0)
  Cycle 2 Day 2, 24 Hours Post-Dose: number analyzed (Participants) | 3 | 10
  Cycle 2 Day 2, 24 Hours Post-Dose | 17.1 (10.4) | 17.2 (7.93)
  Cycle 2 Day 3, 48 Hours Post-Dose: number analyzed (Participants) | 3 | 31
  Cycle 2 Day 3, 48 Hours Post-Dose | 9.60 (5.39) | 16.0 (6.73)
  Cycle 2 Day 3, 96 Hours Post-Dose: number analyzed (Participants) | 3 | 30
  Cycle 2 Day 3, 96 Hours Post-Dose | 6.43 (3.69) | 10.2 (5.16)
  Cycle 3 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 26
  Cycle 3 Day 1, Pre-Dose | 0.415 (0.586) | 1.62 (1.07)
  Cycle 3 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 26
  Cycle 3 Day 1, 5 minutes Post-Dose | 30.0 (5.87) | 38.2 (13.1)
  Cycle 4 Day 1, Pre-dose: number analyzed (Participants) | 2 | 21
  Cycle 4 Day 1, Pre-dose | 0.875 (1.03) | 1.95 (1.26)
  Cycle 4 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 21
  Cycle 4 Day 1, 5 minutes Post-Dose | 29.6 (8.13) | 37.1 (15.6)
  Cycle 5 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 21
  Cycle 5 Day 1, Pre-Dose | 0.844 (0.928) | 2.45 (1.68)
  Cycle 5 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 21
  Cycle 5 Day 1, 5 minutes Post-Dose | 29.4 (3.04) | 38.0 (18.8)
  Cycle 6 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 17
  Cycle 6 Day 1, Pre-Dose | 1.05 (1.20) | 2.99 (1.81)
  Cycle 6 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 17
  Cycle 6 Day 1, 5 minutes Post-Dose | 29.4 (5.37) | 39.8 (19.8)
  Cycle 7 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 17
  Cycle 7 Day 1, Pre-Dose | 0.995 (0.998) | 2.92 (1.62)
  Cycle 7 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 17
  Cycle 7 Day 1, 5 minutes Post-Dose | 24.0 (2.69) | 41.0 (21.2)
  Cycle 8 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 14
  Cycle 8 Day 1, Pre-Dose |  | 3.29 (1.14)
  Cycle 8 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 14
  Cycle 8 Day 1, 5 minutes Post-Dose |  | 41.4 (9.47)
  Cycle 8 Day 2, 24 Hours Post-Dose: number analyzed (Participants) | 0 | 14
  Cycle 8 Day 2, 24 Hours Post-Dose |  | 28.2 (6.38)
  Cycle 8 Day 3, 48 Hours Post-Dose: number analyzed (Participants) | 0 | 14
  Cycle 8 Day 3, 48 Hours Post-Dose |  | 22.9 (5.67)
  Cycle 8 Day 5, 96 Hours Post-Dose: number analyzed (Participants) | 0 | 14
  Cycle 8 Day 5, 96 Hours Post-Dose |  | 17.3 (4.93)
  Cycle 8 Day 14, 312 Hours Post-Dose: number analyzed (Participants) | 0 | 13
  Cycle 8 Day 14, 312 Hours Post-Dose |  | 5.74 (2.02)
  Cycle 9 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 14
  Cycle 9 Day 1, Pre-Dose |  | 6.30 (12.0)
  Cycle 9 Day 1, 5 Minutes Post-Dose: number analyzed (Participants) | 0 | 13
  Cycle 9 Day 1, 5 Minutes Post-Dose |  | 35.1 (11.3)
  Cycle 10 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 12
  Cycle 10 Day 1, Pre-Dose |  | 3.48 (1.13)
  Cycle 10 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 12
  Cycle 10 Day 1, 5 minutes Post-Dose |  | 41.4 (8.63)
  Cycle 11 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 8
  Cycle 11 Day 1, Pre-Dose |  | 3.96 (2.24)
  Cycle 11 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 8
  Cycle 11 Day 1, 5 minutes Post-Dose |  | 42.8 (8.85)
  Cycle 12 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 12 Day 1, Pre-Dose |  | 3.47 (1.28)
  Cycle 12 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 6
  Cycle 12 Day 1, 5 minutes Post-Dose |  | 44.8 (10.3)
  Cycle 13 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 13 Day 1, Pre-Dose |  | 11.3 (17.1)
  Cycle 13 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 3 | 32
  Cycle 13 Day 1, 5 minutes Post-Dose | NA (NA) — No participant was analyzed in this arm group at this time point. | 40.3 (19.2)
  Cycle 14 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 14 Day 1, Pre-Dose |  | 3.97 (1.14)
  Cycle 14 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 6
  Cycle 14 Day 1, 5 minutes Post-Dose |  | 44.5 (7.05)
  Cycle 15 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 15 Day 1, Pre-Dose |  | 4.02 (1.40)
  Cycle 15 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 6
  Cycle 15 Day 1, 5 minutes Post-Dose |  | 49.7 (6.88)
  Cycle 16 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 16 Day 1, Pre-Dose |  | 4.60 (1.67)
  Cycle 16 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 6
  Cycle 16 Day 1, 5 minutes Post-Dose |  | 49.7 (7.61)

21. Secondary Outcome: Monomethyl Auristatin E (MMAE) Plasma Concentrations (Phase 1 and 2)
Description: Blood samples were collected and tested for MMAE plasma concentrations.
Time Frame: as for outcome 4
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1
Number analyzed (Participants) | 3 | 33
ng/mL
  Cycle 1 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 32
  Cycle 1 Day 1, Pre-Dose | NA (NA) — Data was below the limit of quantification. | NA (NA) — Data was below the limit of quantification.
  Cycle 1 Day 1, 5 Minutes Post-Dose: number analyzed (Participants) | 3 | 32
  Cycle 1 Day 1, 5 Minutes Post-Dose | 0.416 (0.480) | 0.368 (0.309)
  Cycle 1 Day 2, 24 Hours Post-Dose: number analyzed (Participants) | 3 | 32
  Cycle 1 Day 2, 24 Hours Post-Dose | 4.63 (3.20) | 4.88 (3.55)
  Cycle 1 Day 3, 48 Hours Post-Dose: number analyzed (Participants) | 3 | 32
  Cycle 1 Day 3, 48 Hours Post-Dose | 4.20 (1.95) | 5.36 (3.72)
  Cycle 1 Day 5, 96 Hours Post-Dose: number analyzed (Participants) | 3 | 32
  Cycle 1 Day 5, 96 Hours Post-Dose | 2.80 (0.300) | 4.43 (3.04)
  Cycle 1 Day 14, 312 Hours Post-Dose: number analyzed (Participants) | 3 | 31
  Cycle 1 Day 14, 312 Hours Post-Dose | 0.196 (0.0641) | 0.530 (0.552)
  Cycle 2 Day 1, Pre-Dose: number analyzed (Participants) | 3 | 29
  Cycle 2 Day 1, Pre-Dose | 0.0647 (0.0358) | 0.0739 (0.0640)
  Cycle 2 Day 1, 5-minutes Post-Dose: number analyzed (Participants) | 3 | 29
  Cycle 2 Day 1, 5-minutes Post-Dose | 0.556 (0.562) | 0.478 (0.461)
  Cycle 2 Day 2, 24 Hours Post-Dose: number analyzed (Participants) | 3 | 8
  Cycle 2 Day 2, 24 Hours Post-Dose | 5.63 (5.72) | 3.71 (3.94)
  Cycle 2 Day 3, 48 Hours Post-Dose: number analyzed (Participants) | 3 | 30
  Cycle 2 Day 3, 48 Hours Post-Dose | 4.60 (3.70) | 3.86 (3.18)
  Cycle 2 Day 5, 96 Hours Post-Dose: number analyzed (Participants) | 3 | 29
  Cycle 2 Day 5, 96 Hours Post-Dose | 2.60 (1.04) | 2.70 (1.69)
  Cycle 3 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 26
  Cycle 3 Day 1, Pre-Dose | 0.0250 (0.0354) | 0.0650 (0.0590)
  Cycle 3 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 25
  Cycle 3 Day 1, 5 minutes Post-Dose | 0.216 (0.0361) | 0.514 (0.684)
  Cycle 4 Day 1, Pre-dose: number analyzed (Participants) | 2 | 19
  Cycle 4 Day 1, Pre-dose | 0.0565 (0.00495) | 0.0866 (0.0784)
  Cycle 4 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 19
  Cycle 4 Day 1, 5 minutes Post-Dose | 0.234 (0.0742) | 0.376 (0.449)
  Cycle 5 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 18
  Cycle 5 Day 1, Pre-Dose | 0.0820 (NA) — Standard deviation was not estimable for 2 participants. | 0.0862 (0.0729)
  Cycle 5 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 18
  Cycle 5 Day 1, 5 minutes Post-Dose | 0.334 (0.0955) | 0.301 (0.248)
  Cycle 6 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 15
  Cycle 6 Day 1, Pre-Dose | 0.0680 (0.0156) | 0.0841 (0.0632)
  Cycle 6 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 15
  Cycle 6 Day 1, 5 minutes Post-Dose | 0.247 (0.00707) | 0.450 (0.663)
  Cycle 7 Day 1, Pre-Dose: number analyzed (Participants) | 2 | 16
  Cycle 7 Day 1, Pre-Dose | 0.104 (0.0389) | 0.0830 (0.0578)
  Cycle 7 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 2 | 15
  Cycle 7 Day 1, 5 minutes Post-Dose | 0.326 (0.0361) | 0.310 (0.282)
  Cycle 8 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 13
  Cycle 8 Day 1, Pre-Dose |  | 0.101 (0.934)
  Cycle 8 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 12
  Cycle 8 Day 1, 5 minutes Post-Dose |  | 0.295 (0.151)
  Cycle 8 Day 2, 24 Hours Post-Dose: number analyzed (Participants) | 0 | 13
  Cycle 8 Day 2, 24 Hours Post-Dose |  | 1.96 (1.31)
  Cycle 8 Day 3, 48 Hours Post-Dose: number analyzed (Participants) | 0 | 13
  Cycle 8 Day 3, 48 Hours Post-Dose |  | 1.91 (1.29)
  Cycle 8 Day 5, 96 Hours Post-Dose: number analyzed (Participants) | 0 | 13
  Cycle 8 Day 5, 96 Hours Post-Dose |  | 2.00 (1.05)
  Cycle 8 Day 14, 312 Hours Post-Dose: number analyzed (Participants) | 0 | 12
  Cycle 8 Day 14, 312 Hours Post-Dose |  | 0.325 (0.214)
  Cycle 9 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 13
  Cycle 9 Day 1, Pre-Dose |  | 0.0819 (0.0496)
  Cycle 9 Day 1, 5 Minutes Post-Dose: number analyzed (Participants) | 0 | 12
  Cycle 9 Day 1, 5 Minutes Post-Dose |  | 0.218 (0.128)
  Cycle 10 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 12
  Cycle 10 Day 1, Pre-Dose |  | 0.727 (0.0517)
  Cycle 10 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 12
  Cycle 10 Day 1, 5 minutes Post-Dose |  | 0.204 (0.0982)
  Cycle 11 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 7
  Cycle 11 Day 1, Pre-Dose |  | 0.0763 (0.0368)
  Cycle 11 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 7
  Cycle 11 Day 1, 5 minutes Post-Dose |  | 0.255 (0.133)
  Cycle 12 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 5
  Cycle 12 Day 1, Pre-Dose |  | 0.105 (0.0983)
  Cycle 12 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 5
  Cycle 12 Day 1, 5 minutes Post-Dose |  | 0.252 (0.116)
  Cycle 13 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 13 Day 1, Pre-Dose |  | 0.110 (0.0629)
  Cycle 13 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 6
  Cycle 13 Day 1, 5 minutes Post-Dose |  | 0.244 (0.130)
  Cycle 14 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 14 Day 1, Pre-Dose |  | 0.109 (0.0529)
  Cycle 14 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 6
  Cycle 14 Day 1, 5 minutes Post-Dose |  | 0.320 (0.138)
  Cycle 15 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 15 Day 1, Pre-Dose |  | 0.0843 (0.0548)
  Cycle 15 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 6
  Cycle 15 Day 1, 5 minutes Post-Dose |  | 0.404 (0.192)
  Cycle 16 Day 1, Pre-Dose: number analyzed (Participants) | 0 | 6
  Cycle 16 Day 1, Pre-Dose |  | 0.139 (0.0926)
  Cycle 16 Day 1, 5 minutes Post-Dose: number analyzed (Participants) | 0 | 6
  Cycle 16 Day 1, 5 minutes Post-Dose |  | 0.381 (0.277)

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after the last dose of study medication (Up to 15 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. At the time of study completion, a total of 9 deaths were reported for the safety population, 1 on study death (death within 30 days of last dose) and 8 deaths during post-treatment follow up (PTFU).
Arm/Group | Brentuximab Vedotin 1.4 mg/kg: Phase 1 | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only
All-Cause Mortality (participants affected / at risk) | 1/3 | 6/16 | 2/17
Serious Adverse Events (participants affected / at risk) | 0/3 | 7/16 | 1/17
Other Adverse Events (participants affected / at risk) | 3/3 | 16/16 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin 1.4 mg/kg: Phase 1 (N=3) | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only (N=16) | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only (N=17)
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with brentuximab 1.8 mg/kg and was not related.
Myalgia (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin 1.4 mg/kg: Phase 1 (N=3) | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r HL Only (N=16) | Brentuximab Vedotin 1.8 mg/kg: Phase 1 and 2 r/r sALCL Only (N=17)
Nausea (Gastrointestinal disorders) | 2 | 7 | 4
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 3
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 8 | 7
Fatigue (General disorders) | 0 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 3 | 4
Pharyngitis (Infections and infestations) | 0 | 3 | 3
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 5 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 3
Migraine (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 4 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 2 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 2 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2014-06-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT01492088/Prot_001.pdf
  • Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT01492088/SAP_000.pdf